CLINICAL TRIAL: NCT07032142
Title: A Phase I/II Trial to Evaluation of the Dose and Efficacy of an Antidote to Fluoropyrimidines
Brief Title: Dose Optimization and Efficacy Assessment of a Fluoropyrimidine Antidote
Acronym: ARCTURUS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Camila Motta Venchiarutti Moniz, Doctor, Principal Investigator, D'Or Institute for Research and Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARCTURUS 81626124.3.1001.5249; 81626124.3.1001.5249 (Other: Regulatory body CEP - CAAE)
Record Dates: First submitted 2025-05-21; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Toxicity Due to Chemotherapy
Keywords: cancer; fluoropyrimidines; Toxicities from Fluoropyrimidines
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who developed severe (grade 3 or higher) toxicities from the use of Fluoropyrimidines (Experimental)
  Interventions: Drug: I-01/23

INTERVENTIONS:
Drug: I-01/23 — The I-01/23 will be administered over a 5-day period, with dosing adjusted according to the patient's body surface area (BSA).

SUMMARY:
Fluoropyrimidines (FLU) are drugs widely used in chemotherapy for various tumors, such as breast, colon, rectal, and gastric cancers. FLU is a drug that inhibits thymine synthesis and, consequently, DNA synthesis, leading to tumor cell death. However, up to 30% of patients treated with FLU experience severe toxicities, depending on the dose and regimen received. The most common symptoms include mucositis, vomiting, nausea, diarrhea, and neutropenia.

The enzyme dihydropyrimidine dehydrogenase (DPD) plays a key role in FLU metabolism. Patients with mutations in the DPYD gene (which encodes DPD) are at high risk of experiencing severe toxicities from FLU. Uridine triacetate (UT) is a drug that can be used as an antidote for 5-FU in patients who develop severe toxicities. However, despite its efficacy, it is expensive and not commercially available in Brazil.

Currently, the Brazilian population has no access to an antidote for the treatment of FLU-related toxicities. This Phase I/II study will evaluate the dose, safety, and efficacy of compound the association of two molecules as an antidote for grade 3 or higher toxicities resulting from the use of FLU.

ELIGIBILITY:
Inclusion Criteria:

Presence of at least one severe toxicity or intoxication resulting from fluoropyrimidine use, defined as: receiving an overdose of medication (total dose and/or infusion rate higher than recommended in the package insert) and/or Grade 3 or 4 serious adverse events after fluoropyrimidine exposure, according to CTCAE v5.0, which may include (but are not limited to): nausea, vomiting, diarrhea, anemia, neutropenia, febrile neutropenia, thrombocytopenia, and mucositis;

Lack of access to uridine triacetate (UT) in the standard of care;

Diagnosis of an invasive solid tumor under systemic treatment with a fluoropyrimidine (5-fluorouracil or capecitabine);

Organ function considered adequate by the investigator prior to the current fluoropyrimidine intoxication episode;

Ability to take oral medication;

For men and women of reproductive potential, agreement to practice abstinence or use highly effective contraceptive methods during study participation and for at least 6 months after the last dose of IP;

Men must agree not to donate sperm for at least 6 months after the last dose of IP;

Body surface area between 1.4 and 2.4 m², calculated using the Du Bois method;

AST/ALT within normal limits for participants without liver metastases;

AST/ALT up to 3x the upper limit of normal in participants with liver metastases;

Total and fractionated bilirubin up to 2x the upper limit of normal;

Agreement to abstain from alcohol consumption during the treatment period;

As a specific inclusion criterion for participants in Phase 1 of the study: a medical indication, according to routine care, for hospitalization of at least 48 hours for the clinical management of fluoropyrimidine-related toxicity.

Exclusion Criteria:

Pregnant or breastfeeding women;

Known history of allergic reaction to the molecules of the copound and/or to other molecules in the same class;

Life expectancy of less than 30 days prior to hospital admission, based on underlying cancer and existing comorbidities;

Estimated creatinine clearance <70 mL/min;

Liver cirrhosis;

Known liver or kidney disease;

Individuals with acquired immunodeficiency may be included only if they have no active opportunistic infections and following careful clinical assessment by the investigator, taking into account concurrent medications;

Family history or known deficiency of the enzyme responsible for metabolizing the molecules of the copound and/or to other molecules in the same class;

Uncontrolled infection;

Hemodynamically unstable patients;

Patients under orotracheal intubation;

Patients unable to take oral medication;

Prolonged QT interval;

CNS metastases considered uncontrolled by the investigator;

History of malabsorptive or inflammatory gastrointestinal disease;

Use within the last 30 days of lactulose, protease inhibitors, amiodarone, carbamazepine, phenytoin, phenobarbital, oxcarbazepine, rifabutin, rifampin, or rifapentine;

Use within the last 5 days of dietary supplements containing the molecules of the copound;

Use within the last 30 days of drugs classified as anticonvulsants;

Personal history of seizures;

Comorbidities deemed limiting by the investigator;

History of renal or liver transplant;

Presence of intestinal obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Determination | 6 days
  Definition of DMT (Phase I) : The maximum tolerated dose (DMT) is the highest dose that produces the desired effect without resulting in unacceptable side effects
Survival rate | 7 days
  The rate will be calculated as the percentage of participants alive following the initiation of treatment

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Instituto D'Or de Pesquisa e Ensino de Salvador, Salvador, Estado de Bahia
  - Instituto D'Or de Pesquisa e Ensino de Brasília, Brasília, Federal District
  - Instituto D'Or de Pesquisa e Ensino de Curitiba, Curitiba, Paraná
  - Instituto D'Or de Pesquisa e Ensino do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No